CLINICAL TRIAL: NCT00277004
Title: Physiological Biomarkers of Cancer Treatment Related Fatigue in Women With Breast Cancer.
Status: Terminated | Type: Observational
Why Stopped: This is not a clinical trial and was entered in the system in error.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: 0399C
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Breast; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Physiological Biomarkers of Cancer Treatment Related Fatigue in Women with Breast Cancer.

DETAILED DESCRIPTION:
As above.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed early stage breast cancer.

Exclusion Criteria:

* Not specified.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Females with breast cancer undergoing cancer treatment.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 1999-02 (Actual); Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Disease Progression | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian Rabinowitz, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States